CLINICAL TRIAL: NCT05400980
Title: The Expander-2 Trial: A Multi-Center, Randomized, Blinded, Controlled Study to Evaluate the Safety and Efficacy of the Urocross® Expander System and Retrieval Sheath
Brief Title: Expander-2 Trial: Randomized Study to Evaluate Safety & Efficacy of the Urocross® Expander System & Retrieval Sheath
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prodeon Medical, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CP002
Record Dates: First submitted 2022-05-27; First posted 2022-06-02 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-01

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Prostate; BPH; Benign; Minimally Invasive; Temporary
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: Randomization in a ratio 2:1 Urocross Expander implant using the Urocross Expander System vs. Sham control (cystoscopy only)
Who Masked: Participant, Outcomes Assessor
Masking Description: All subjects will be blinded to the treatment assignment up to the primary efficacy endpoint (3 months post-procedure).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Urocross implant group (Experimental): The investigational products in this trial are the Urocross Expander Implant as delivered by the Urocross Expander System and the Urocross Retrieval Sheath used to retrieve the implant after 6 months following its implant.
  Interventions: Device: Urocross implant
- Sham-control group (Sham Comparator): The sham-control in this trial is cystoscopy only.
  Interventions: Diagnostic Test: Sham-control

INTERVENTIONS:
Device: Urocross implant — Urocross implant inserted via delivery catheter
  Arms: Urocross implant group
Diagnostic Test: Sham-control — Cystoscopy
  Arms: Sham-control group

SUMMARY:
To demonstrate the safety and efficacy of the Urocross Expander System/Retrieval Sheath and the procedure to treat patients with symptomatic Benign Prostatic Hyperplasia (BPH).

DETAILED DESCRIPTION:
Pivotal, prospective, multi-center, randomized, sham-controlled, blinded study

ELIGIBILITY:
Inclusion Criteria:

1. Subject has signed an informed consent form (ICF).
2. Men ≥ 45 years.
3. Symptomatic BPH with the following (all must be met):

   * IPSS ≥ 13.
   * Qmax ≤ 12 mL/sec on a voided volume of ≥ 125 mL.
   * PVR < 250 mL.
4. Prostate volume 30-80 cc measured by transrectal ultrasound (TRUS) or magnetic resonance imaging (MRI) within 6 months prior to randomization.
5. Subjects willing to be off their BPH-related medications from time of enrollment and throughout study participation.

Note: All subjects on BPH-related medications must start a washout period prior to qualifying questionnaires and uroflowmetry.

Exclusion Criteria:

Subjects who meet ANY of the following exclusion criteria will not participate in the trial:

1. Previous BPH procedure intended to disobstruct the bladder outlet (e.g., prostate surgery, stent implantations, laser prostatectomy, hyperthermia or another invasive treatment to the prostate).
2. Obstructive protruding (mobile) middle (median) prostatic lobe as confirmed by cystoscopy.
3. High bladder neck as determined by the Investigator.
4. Urethral stricture, meatal stenosis, or bladder neck contraction - either current, or recurrent requiring 2 or more dilatations.
5. Biopsy of the prostate within past 8 weeks.
6. Baseline Prostate Specific Antigen (PSA) level > 10 ng/mL or confirmed or suspected prostate cancer (subjects with a PSA level > 2.5 ng/mL or whose PSA levels fall outside age-specific or local reference ranges, should have prostate cancer excluded to the Investigator's satisfaction in conjunction with shared decision making [SDM] with the study subjects).
7. Confirmed or suspected bladder cancer.
8. History of cystolithiasis, kidney stone, or kidney disease within the prior 3 months.
9. History of neurogenic bladder.
10. Previous episode of AUR, i.e., post hernia repair or other condition or disease that might cause urinary retention.
11. Parkinson's disease or other neurologic disease known to impact bladder function (e.g., stroke, TIA, multiple sclerosis).
12. Serum creatinine > 1.8 mg/dL or renal dysfunction attributed to bladder outlet obstruction (BOO).
13. Concomitant UTI (subject can be enrolled following successful treatment of UTI and a negative UTI test), or subjects who have a history of recurrent or chronic UTIs (defined as 2 or more UTIs in the past 12 months).
14. Active infection including acute bacterial prostatitis.
15. Previous pelvic irradiation or radical pelvic surgery.
16. Known allergy to nickel.
17. Subjects with life-threatening disease in which life expectancy is foreshortened are excluded.
18. Desire to maintain fertility post-treatment.
19. Anticipated need for additional major surgery or treatments for comorbidities during the study period (e.g., valve repair, organ transplant).
20. Prostatic urethral length < 25 mm or > 60 mm, as measured from bladder neck to verumontanum, using cystoscopy just prior to randomization.
21. Any concurrent medical condition or illness that might prevent study completion or that could impact the study results such as:

    * severe cardiac arrhythmias uncontrolled by medications or pacemaker.
    * congestive heart failure New York Heart Association (NYHA) III or IV.
    * uncontrolled diabetes mellitus.
    * significant respiratory disease in which hospitalization may be required.
    * known immunosuppression (i.e., AIDS, post-transplant, undergoing chemotherapy).
22. Inability to stop taking anticoagulants and/or antiplatelets for at least 3 days prior to the procedure or coumadin for at least 5 days prior to the procedure.

    Note: Low dose aspirin therapy is acceptable.
23. Unable or unwilling to complete all required questionnaires and follow-up assessments.
24. Participating in any other investigational study for either drug or device which can influence collection of valid data under this study.
25. Subject is in custody or institution, or, in the Investigator's opinion, has a physical, psychological, or medical impairment that might prevent study completion or would confound study results (including subject questionnaires).

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Safety of Urocross Expander Implant | more than 7 days post procedure
  The rate of extended post-operative urinary catheterization (more than 7 days) from treatment for inability to void.
Efficacy of the Urocross Expander Implant as delivered by the Urocross Expander System and the Urocross Retrieval Sheath | 3 months post-procedure
  The primary efficacy endpoint is Change from Baseline in Total International Prostate Symptom Score (IPSS) at 3 months post-procedure. The IPSS items range in score from 0-5, with higher scores indicating worse symptoms. The study is powered to show that the average improvement in Total IPSS among the Urocross Implant subjects is more than 25% greater than the average improvement in Total IPSS among the sham-control subjects.

SECONDARY OUTCOMES:
Percent change in Total IPSS for subjects randomized to the Urocross Implant | 3 months post-procedure
  The major secondary efficacy endpoint is the percent change in Total IPSS from baseline (i.e., pre-procedure) to 3 months post-procedure for subjects randomized to the Urocross Implant group. The IPSS items range in score from 0-5, with higher scores indicating worse symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin T. McVary, Principal Investigator — Loyola University; Daniel B. Rukstalis, Principal Investigator — Carilion Clinic
Locations (2):
- United States (2):
  - Loyola University Medical Center, Maywood, Illinois
  - Virginia Tech-Carilion School of Medicine, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No